CLINICAL TRIAL: NCT06170528
Title: ARUA-ALZ - Connecting Audio and Radio Sensing Systems to Improve Care at Home for ADRD
Brief Title: ARUA-ALZ - Connecting Audio and Radio SensingmSystems to Improve Care at Home for ADRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Jing Wang, FSU Site Principal Investigator, Florida State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00003184
Record Dates: First submitted 2023-10-19; First posted 2023-12-14 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer Disease; Caregiver Burden
MeSH Terms: conditions — Alzheimer Disease; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Mild ADRA and their caregivers (Other): Deployed the AURA_ALZ system at Home
  Interventions: Device: AURA_ALZ

INTERVENTIONS:
Device: AURA_ALZ — AURA_ALZ includes the WiFi CSI-based human sensing algorithms, as well as the voice and web interfaces. The devices of AURA_ALZ consists of Fitbit watch, iPad, ASUS routers, Jetson nano, webcam, and Amazon Echo.

SUMMARY:
The purpose of this study is to address the unmet care needs and reduce the care burdens for persons with ADRD (Alzheimer's Disease and Alzheimer's Disease Related Dementias) and their caregivers by providing monitoring of daily activities and gestures using audio and radio sensing, providing voice-based reminders intervention.

In phase 1, dyads will participate in two focus groups will take 60 minutes per each. In Phase 2, AURA_ALZ (connecting Audio and Radio Sensing Systems-Alzheimer's Disease) will deployed for two weeks at participants' home. At the end of the two weeks, usability, acceptability of the use of the system will be measured.

DETAILED DESCRIPTION:
The purpose of this study is to reduce the care burdens of people with mild cognitive impairment or mild dementia and their caregivers using Fitbit watches and Amazon Echo devices. Couples will be both recruited and provided with consent forms that explain the study.

In the first phase, after the informed consent, selected dyads will participate in two focus groups will take 60 minutes per each. For this, a research staff will schedule a zoom meeting and then will show the short introduction video regarding Alexa and Fitbit, lists of voice interaction with Alexa, and lists of Fitbit conversation. After this, each dyad will participate in one focus groups interview.

In the second phase, a researcher will visit each dyad's home to set up Amazon Echo and Fitbit. The research staff will train participants in use of the Amazon Echo device and Fitbit. A web camera will be set up in the living room. This visit will take about three hours. The camera will run for three hours, and then be removed from the home setting. Two routers, the Amazon echo, Fitbit watch and iPad will remain in the home for two weeks. Signals from two routers will capture activities. Couples will contact the researcher with questions. During the two weeks data on movement, sitting, lying, walking, drinking, eating, falls, washing face, brushing teeth, and location data of the patients as detected by the WIFI router. Daily reminders will be given through the voice assisted ECHO system for routine activities of daily living including time to eat, taking medication, etc. At the end of the two-week study period, measurements will be made on usability, acceptability of the use of the system. Participants will be compensated with another $50.00 gift card for completing this phase of the study.

There are minimal risks in performing the research procedures that consist of a survey, interview, and testing feasibility of the device. However, PI will continuously monitor any harms or discomfort from participants.

Data reporting: Information the investigators learn about participants in this study will be handled in a confidential manner, within the limits of the law. If investigators publish the results of the study in a scientific journal or book, no participants will be identified. The Institutional Review Board and other groups that have the responsibility of monitoring research may want to see study records which identify the participants as a subject in this study.

ELIGIBILITY:
Inclusion Criteria:

* To be included, dyads of persons with ADRD and their family caregivers must meet the following criteria:

  1. 1 person must be diagnosed with ADRD from a physician. Caregivers must self-report that their person's dementia diagnosis from a physician and self-report Global Deterioration Scale (GDS) rating for care recipients to determine stage of dementia. Eligible participants must characterize their person's ADRD symptoms as fitting with Stages 3 and 4 (defined as mild cognitive impairment to mild dementia of Alzheimer's type),
  2. at least 1 caregiver living in the same household for at least 4 hours per day for at least the past 6 months,
  3. both individuals within the dyads be at least 18 years of age,
  4. both individuals within the dyads have sufficient vision and speaking capabilities to use a voice-enabled system, and
  5. both individuals within the dyads live in a community setting in Tallahassee or assisted living setting inTallahassee.

Exclusion Criteria,

1. Person is diagnosed with Moderate and Sever ADRD
2. No caregivers living in the same household
3. Both individuals with less 18 years of age
4. Both individuals within the dyads have language barriers

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Usability of use of the AURA_ALZ system will be determined | At two weeks after deployment of system
  Usability Scale (rating from 1 to 5 with the higher score is better)adapted for the evaluation of AURA-ALZ will be administered to assess the usability of AURA-ALZ.
Acceptability of use of the AURA_ALZ system will be determined | At two weeks after deployment of system
  Interviews will be conducted with all study participants to ask about their acceptability of the AURA-ALZ system
Feasibility of use of the AURA_ALZ system will be determined | At two weeks after deployment of system
  Feasibility will be determined by the retention rates.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wang, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University College of nursing, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No